CLINICAL TRIAL: NCT00522067
Title: A Phase II, Open Label, Uncontrolled, Multi-Center Study to Support Annual Strain Update and to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Adjuvanted Influenza Vaccine, Formulation 2007-2008, When Administered to Subjects Aged 18-64 Years Affected by Chronic Diseases
Brief Title: Support Annual Strain Update, Safety and Immunogenicity of an Inactivated, Adjuvanted Influenza Vaccine, Formulation 2007-2008, When Administered to Subjects 18-64 Years Affected by Chronic Diseases.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70P4; 2007-000964-26
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-01

CONDITIONS: Influenza Disease
Keywords: influenza; influenza vaccine; adjuvanted influenza vaccine; subunit influenza vaccine; surface antigen
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): FLUAD
  Interventions: Biological: Adjuvanted influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted influenza vaccine — Vaccination with MF 59 adjuvanted trivalent seasonal influenza vaccine

SUMMARY:
This phase II, open label, is designed as a seasonal study to support annual strain update evaluating the safety, clinical tolerability and immunogenicity of the 2007-2008 formulation of Novartis Vaccines' adjuvanted, subunit influenza vaccine in adults with underlying chronic diseases

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years of age adult volunteers, mentally competent, willing and able to give written informed consent prior to study entry, suffering from at least one of these chronic diseases: hypertension, heart disease, chronic obstructive pulmonary disease (COPD) or asthma, hepatic or renal insufficiency, arteriosclerotic disease or insulin dependent diabetes mellitus

Exclusion Criteria:

* Hypersensitivity to ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate or any other component of the vaccine;
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
* Known or suspected impairment/ alteration of immune function;
* Having received within the past 12 months more than one injection of influenza vaccine
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the antibody response to each flu vacc. antigen, measured by SRH at 21-day post-vacc. in at risk adults in compliance with the requirements of the EU recommendations for the evaluation of the immunog. for a new formulation of a licensed flu vacc
To evaluate the safety of the administration of a single intramuscular(IM) injection of an inactivated, adjuvanted influenza vaccine, in at risk adult subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Azienda Sanitaria USL 7 di Siena, Siena, Italy